CLINICAL TRIAL: NCT05803967
Title: Baduanjin Exercising Effects on Women With Hypothyroidism and Cognitive Problems
Brief Title: Baduanjin Exercising Effects on Sub-clinical Hypothyroidism and Cognitive Problems
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ali Mohamed Ali ismail, lecturer of physical therapy for Internal Medicine and Geriatrics, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004294
Record Dates: First submitted 2023-03-27; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Subclinical hypothyroïdism; Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group number 1 (Experimental): Females with sub-clinical hypothyroidism exhibit cognitive problems (mild cognitive impairement), they will be elderly, will receive baduanjin training that will be applied 5 times per the week, under supervision for 12 weeks, number of patients will be 20), also women of this group will receive their prescribed daily one-dose medication tablet (levothyroxine).
  Interventions: Behavioral: Baduanjin exercising
- group number 2 (No Intervention): Females with sub-clinical hypothyroidism exhibit cognitive problems (mild cognitive impairement), they will be elderly, will receive will receive their prescribed daily one-dose medication tablet (levothyroxine).

INTERVENTIONS:
Behavioral: Baduanjin exercising — baduanjin will be applied 5 times per the week, under supervision, for 12 weeks,
  Arms: group number 1

SUMMARY:
Females with sub-clinical hypothyroidism may exhibit frequent cognitive problems especially if they are elderly

DETAILED DESCRIPTION:
Females (forty in number) with sub-clinical hypothyroidism exhibit cognitive problems, they are elderly, will be divided to exercised group (baduanjin training will be applied 5 times per the week, under supervision for 12 weeks, number of patients will be 20) and other non exercised group (number of patients will be 20) . all women of groups will received their prescribed daily one-dose medication tablet (levothyroxine).

ELIGIBILITY:
Inclusion Criteria:

* female with sub-clinical hypothyroidism
* females with mild cognitive impairment
* females with obesity (obesity class one)

Exclusion Criteria:

* neurological problems
* orthopedic problems

Ages: 65 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Older Adult
Gender Based: Yes — based on self-representation of gender identity.
Enrollment: 40 (Estimated)
Dates: Start 2022-12-18 (Actual); Primary Completion 2023-06-18 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
thyroid stimulating hormone | it will be measured after 12 weeks
  will be measured in serum of women with hypothyroidism

SECONDARY OUTCOMES:
systolic blood pressure | it will be measured after 12 weeks
  will be measured by manual sphygmomanometer
triglycerides | it will be measured after 12 weeks
  will be measured in serum of women with hypothyroidism
Addenbrooke Cognitive Examination | it will be measured after 12 weeks
  will assess Cognitive impairment
diastolic blood pressure | it will be measured after 12 weeks
  will be measured by manual sphygmomanometer
low density lipoprotein | it will be measured after 12 weeks
  will be measured in serum of women with hypothyroidism
cholesterol | it will be measured after 12 weeks
  will be measured in serum of women with hypothyroidism
high density lipoprotein | it will be measured after 12 weeks
  will be measured in serum of women with hypothyroidism
body mass index | it will be measured after 12 weeks
  it will be measure on empty bladder and stomach

CONTACTS AND LOCATIONS:
Overall Officials: Ali MA Ismail, Principal Investigator — Cairo University
Locations (1):
- Cairo Unoversity, Giza, Egypt